CLINICAL TRIAL: NCT06370429
Title: The Effect of Progressive Relaxation Exercises Performed Online by Women With Premenstrual Syndrome on the Stress Level and Family Functionality of Women and Their Spouses
Brief Title: Effect of Online Exercises for Premenstrual Syndrome on Couple's Stress and Family Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ayşe Sevim AKBAY KISA, research assistant, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 8743432956-050.99-621064
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Premenstrual Syndrome; Exercises; Stress Level; Family Characteristics
Keywords: Premenstrual Syndrome; Progressive Relaxation; Stress Level; Family Functionality
MeSH Terms: conditions — Premenstrual Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: The sample was divided into intervention and control groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Relaxation Exercises (Experimental): Progressive Relaxation Exercises, randomized pretest-posttest
  Interventions: Other: Progressive Relaxation Exercises, randomized pretest-posttest
- control (No Intervention): Non-intervention

INTERVENTIONS:
Other: Progressive Relaxation Exercises, randomized pretest-posttest — experimental and control ,a randomized pretest-posttest study to examine
  Arms: Progressive Relaxation Exercises

SUMMARY:
Universe of Research The universe of the research; It will consist of women and their spouses with premenstrual syndrome complaints who use social media.

3.6. Sample of the Research The number of samples of the study was composed of a total of 60 (Intervention = 30, Control = 30) participants.

Criteria for inclusion in the study:

* Being married and living with his wife
* Being between the ages of 18-45,
* The woman's ability to use a mobile phone and/or computer to receive online
* The woman and her husband must be literate
* The woman does not have a hearing problem that would prevent her from understanding the voice recording, 9. Scoring 110 or above on the Premenstrual Syndrome Scale 10. Having regular menstrual cycles for the last six months, 13. Having no other medical disease in the last six months, 14. Participant who does not use oral contraceptives, 16. Not pregnant or breastfeeding, 17. No history of cancer. 18. Those who do not use medical drugs to reduce premenstrual syndrome 19. Those who do not use herbal medicine to reduce premenstrual syndrome 20. Do not practice exercise, yoga, etc. to reduce premenstrual syndrome.

Exclusion criteria from the study:

1. He or his spouse fills out the research survey forms incompletely,
2. Pregnancy occurs,
3. Receiving breathing exercise consultancy from another consultant during the study period

Data Collection Method and Duration Descriptive Characteristics Data Form, Perceived Stress Scale (PSS) and Family Assessment Scale will be applied to the sampled women and their spouses. Data collection will continue until the calculated sample number is reached.

DETAILED DESCRIPTION:
Type of research The research will be conducted as a randomized controlled intervention study to Examine the Effects of Progressive Relaxation Exercises Performed Online by Women with Premenstrual Syndrome on the Stress Level and Family Functionality of Women and Their Spouses.

Universe of Research The universe of the research; It will consist of women and their spouses with premenstrual syndrome complaints who use social media.

3.6. Sample of the Research The sample of the research will consist of women who meet the inclusion criteria. The number of samples was calculated by the researchers using the Power analysis Power 3.1 package program. The sample calculation was based on the study titled 'The Effect of Progressive Relaxation Exercises on Stress Level, Sleep Quality and Exercise Capacity in Young Adults' in the pre-pandemic period in Turkish culture. 80% power from the study of Oğuz et al (2019); By calculating the sample size at an effect size of 0.82 and an error level of 0.05, it was determined that 20 women each should be included in the intervention and control groups in the study. However, since spouses will also participate in the survey process, considering that there may be losses for women and their spouses, the number of participants in each group was increased by 50% and the sample of the study was composed of a total of 60 (Intervention = 30, Control = 30) participants.

Criteria for inclusion in the study:

1. Volunteering to participate in the study, 2. Being married and living with his wife 3. Being between the ages of 18-45, 5. The woman's ability to use a mobile phone and/or computer to receive online (Zoom; social media) counseling and listen to exercises, 6. The woman and her husband have a social media., application or e-mail address.

7. The woman and her husband must be literate 8. The woman does not have a hearing problem that would prevent her from understanding the voice recording, 9. Scoring 110 or above on the Premenstrual Syndrome Scale 10. Having regular menstrual cycles for the last six months, 11. Not having undergone bilateral oophorectomy or hysterectomy, 12. Not having been diagnosed with polycystic ovary syndrome, 13. Having no other medical disease in the last six months, 14. Participant who does not use oral contraceptives, 15. Without severe psychosomatic disorder, 16. Not pregnant or breastfeeding, 17. No history of cancer. 18. Those who do not use medical drugs to reduce premenstrual syndrome 19. Those who do not use herbal medicine to reduce premenstrual syndrome 20. Do not practice exercise, yoga, etc. to reduce premenstrual syndrome.

Exclusion criteria from the study:

1. He or his spouse fills out the research survey forms incompletely,
2. Wanting to leave the research at any stage of the research,
3. Not participating in the final test,
4. Pregnancy occurs,
5. Receiving breathing exercise consultancy from another consultant during the study period
6. Those who do the relaxation exercises incorrectly according to the Content of the Progressive Relaxation Exercises,

Data Collection Method and Duration Descriptive Characteristics Data Form, Perceived Stress Scale (PSS) and Family Assessment Scale will be applied to the sampled women and their spouses. Data collection will continue until the calculated sample number is reached.

Hypotheses:

H1: There is a difference between the mean stress level scores of women with premenstrual syndrome who take online progressive relaxation exercises and women who do not.

H2: There is a difference between the mean stress level scores of women with premenstrual syndrome who receive online progressive relaxation exercises and the spouses of women who do not.

H3: There is a difference between the mean family functionality score of women with premenstrual syndrome who receive online progressive relaxation exercises and those who do not.

H4: There is a difference between the mean family functionality scores of women with premenstrual syndrome who receive online progressive relaxation exercises and their spouses who do not.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study,
2. Being married and living with his wife
3. Being between the ages of 18-45,
4. The woman's ability to use a mobile phone and/or computer to receive online (Zoom; vs) counseling and listen to exercises,
5. The woman and her husband have a application or e-mail address that can use the googledocs application.
6. The woman and her husband must be literate
7. The woman does not have a hearing problem that would prevent her from understanding the voice recording,
8. Scoring 110 or above on the Premenstrual Syndrome Scale
9. Having regular menstrual cycles for the last six months,
10. Not having undergone bilateral oophorectomy or hysterectomy,
11. Not having been diagnosed with polycystic ovary syndrome,
12. Having no other medical disease in the last six months,
13. Participant who does not use oral contraceptives,
14. Without severe psychosomatic disorder,
15. Not pregnant or breastfeeding,
16. No history of cancer.
17. Those who do not use medical drugs to reduce premenstrual syndrome
18. Those who do not use herbal medicine to reduce premenstrual syndrome
19. Do not practice exercise, yoga, etc. to reduce premenstrual syndrome.

Exclusion Criteria:

1. He or his spouse fills out the research survey forms incompletely,
2. Wanting to leave the research at any stage of the research,
3. Not participating in the final test,
4. Pregnancy occurs,
5. Receiving breathing exercise consultancy from another consultant during the study period
6. Those who do the relaxation exercises incorrectly according to the Content of the Progressive Relaxation Exercises CD,

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale | The research period for a participant takes approximately 3 months.
  It is a 44-item, five-point Likert-type scale (Never, Very little, Sometimes, Frequently, Continuously) developed by Gencdogan and measures the severity of premenstrual symptoms.
  In scoring the scale, the "Never" option is evaluated as 1 point, the "Very little" option is evaluated as 2 points, the "Sometimes" option is evaluated as 3 points, the "Often" option is evaluated as 4 points and the "Always" option is evaluated as 5 points.
  The lowest score that can be obtained from the scale is 44 and the highest score is 220. The higher the score, the more intense the premenstrual syndrome symptoms are considered.
Family Assessment Scale | The research period for a participant takes approximately four months.
  Its original form was developed by Brown University and Butler Hospital in the United States within the framework of the Family Research Program. The family evaluation scale consists of 60 (sixty) questions and 7 sub-dimensions. It is a scale with four options and each item is scored between 1.00 (healthy) and 4.00 (unhealthy). Minimum 60 and maximum 240 points are taken from the scale. As the score increases, it indicates that family functionality is not good.
Perceived Stress Scale | The research period for a participant takes approximately four months.
  Perceived Stress Scale (PSS) Cohen consists of 14 items in total. The scale is a five-point Likert type in which each item is scored between "Never (0)" and "Very often (4)". The total score obtained from the scale ranges from 0 to 56, and the score obtained from 11 to 26 is considered low; 27-41 is medium; 42-56 indicates high stress level.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba NU KORKMAZ ASLAN, Study Chair — Necmettin Erbakan University; Gazi ÇU Kısa, Study Chair — Cukurova University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No